CLINICAL TRIAL: NCT03225352
Title: An Open Label, Randomized, Four-Way Crossover Trial to Assess the Disintegration, Gastric Emptying and Pharmacokinetic Parameters of a New Disintegrating Acetylsalicylic Acid 500 mg, 1000 mg Tablet Formulation and 2 Different Ibuprofen Tablets in Fasted Healthy Male Subjects
Brief Title: A Study to Assess Disintegration of the New Aspirin Disintegrating Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19220; 2016-004546-29 (EudraCT Number)
Record Dates: First submitted 2017-07-16; First posted 2017-07-21 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Moderate Pain
MeSH Terms: interventions — Aspirin; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1: starting with BAYE4465 500 mg (Experimental): Participants will participant four treatment periods with four different treatments. Treatment assignment adhere to Williams design
  Interventions: Drug: 500 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 1000 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 400 mg ibuprofen(Nurofen); Drug: 400 mg ibuprofen (Dolormin Extra)
- Sequence 2: starting with BAYE4465 1000 mg (Experimental): Participants will participant four treatment periods with four different treatments. Treatment assignment adhere to Williams design
  Interventions: Drug: 500 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 1000 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 400 mg ibuprofen(Nurofen); Drug: 400 mg ibuprofen (Dolormin Extra)
- Sequence 3: starting with Nurofen (Experimental): Participants will participant four treatment periods with four different treatments. Treatment assignment adhere to Williams design
  Interventions: Drug: 500 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 1000 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 400 mg ibuprofen(Nurofen); Drug: 400 mg ibuprofen (Dolormin Extra)
- Sequence 4: starting with Dolormin Extra (Experimental): Participants will participant four treatment periods with four different treatments. Treatment assignment adhere to Williams design
  Interventions: Drug: 500 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 1000 mg acetylsalicylic acid (Aspirin, BAYE4465); Drug: 400 mg ibuprofen(Nurofen); Drug: 400 mg ibuprofen (Dolormin Extra)

INTERVENTIONS:
Drug: 500 mg acetylsalicylic acid (Aspirin, BAYE4465) — Single intake of 1 tablet, 500mg
Drug: 1000 mg acetylsalicylic acid (Aspirin, BAYE4465) — Single intake of 1 tablet, 1000mg
Drug: 400 mg ibuprofen(Nurofen) — Single intake of 1 tablet, 400mg
Drug: 400 mg ibuprofen (Dolormin Extra) — Single intake of 1 tablet, 400mg

SUMMARY:
The aim of this study is to assess disintegration of the new Aspirin disintegrating tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 65 years included
* Verified diagnosis of "healthy"
* Non-smokers or passive smokers
* BMI in the range of 18.5 to 30 kg/m2
* Subject has given written informed consent to participate in the trial prior to admission to the trial

Exclusion Criteria:

* Blood donation within the last 90 days prior to planned randomization
* Any previous medication within 10 days before the planned administration of the radiolabelled Investigational Medicinal Product (rIMP) which, in the opinion of the physician responsible, will interfere with the study procedures or compromise safety
* Subject has any non-removable metal objects such as metal plates, screws etc. in their chest or abdominal area which, in the opinion of the physician responsible, could affect the study conduct.
* Vegetarian
* Subjects for whom participation in this study will exceed the limits of total radiation exposure allowed in any 12 month period (5 Millisievert), or will exceed 10 Millisievert over any three year period

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Time to complete tablet disintegration | Up to 4 hours
  The tablet is radiolabeled. Scintigraphy images of the abdominal area will be taken It is time until an image with no definable hot spot remaining is identified

SECONDARY OUTCOMES:
Gastric empty time, if applicable | Up to 4 hours
  Gastric emptying time will be calculated by a qualified assessor based on the scintigraphy images
Time of colon arrival, if applicable | Up to 4 hours
  Time of colon arrival will be calculated by a qualified assessor based on the scintigraphy images
Small intestine transit time, if applicable | Up to 4 hours
  Small intestine transit time will be calculated by a qualified assessor based on the scintigraphy images
Time of onset of release of radiolabel | Up to 4 hours
  Time of onset of release of radiolabel will be calculated by a qualified assessor based on the scintigraphy images
Site of onset of release of radiolabel | Up to 4 hours
  Site of onset of release of radiolabel will be determined by a qualified assessor based on the scintigraphy images
Site of completion of release of radiolabel | Up to 4 hours
  Site of completion of release of radiolabel will be determined by a qualified assessor based on the scintigraphy images
Disintegration rate of the tablet estimated from the radioactivity remaining | Up to 4 hours
  Disintegration rate of the tablet estimated from the radioactivity rem will be calculated by a qualified assessor based on the scintigraphy images
Time of 50% disintegration of the tablet estimated from the radioactivity remaining | Up to 4 hours
  Time of 50% disintegration of the tablet estimated from the radioactivity remaining will be calculated by a qualified assessor based on the scintigraphy images
Gastric emptying kinetics of dispersed radioactive material (t50% and t90%) | Up to 4 hours
  Gastric emptying kinetics of dispersed radioactive material (t50% and t90%) will be calculated by a qualified assessor based on the scintigraphy images
AUC0-t | Prior to dosing (between 60-15 min), and 5, 9, 13, 18, 23, 28, 33, 38, 48, 58, 68, 78, 88, 118, 178 and 238 min post-dose
  Area under the plasma concentration vs time curve from zero to the last data point
Cmax | Prior to dosing (between 60-15 min), and 5, 9, 13, 18, 23, 28, 33, 38, 48, 58, 68, 78, 88, 118, 178 and 238 min post-dose
  Maximum drug concentration in plasma after single dose administration
AUC0-infinity | Prior to dosing (between 60-15 min), and 5, 9, 13, 18, 23, 28, 33, 38, 48, 58, 68, 78, 88, 118, 178 and 238 min post-dose
  Area under the plasma concentration vs time curve from zero to infinity
t1/2 | Prior to dosing (between 60-15 min), and 5, 9, 13, 18, 23, 28, 33, 38, 48, 58, 68, 78, 88, 118, 178 and 238 min post-dose
  Half-life associated with the terminal slope
tmax | Prior to dosing (between 60-15 min), and 5, 9, 13, 18, 23, 28, 33, 38, 48, 58, 68, 78, 88, 118, 178 and 238 min post-dose
  Time to reach maximum drug concentration in the measured
Cmax/AUC0-infinity | Prior to dosing (between 60-15 min), and 5, 9, 13, 18, 23, 28, 33, 38, 48, 58, 68, 78, 88, 118, 178 and 238 min post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-Images Research Ltd, Glasgow, Glasgow City, United Kingdom